CLINICAL TRIAL: NCT03358342
Title: ePneumonia: Development of an Electronic Clinical Decision Support System for Community-Onset Pneumonia
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Nathan Dean, Section Chief of Pulmonary and Critical Care Medicine, Intermountain Health Care, Inc.
Other Study IDs: ePneumonia - CDS
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ED Patients treated using ePneumonia CDS: ED patients with community-acquired pneumonia treated in ED's after roll out of ePneumonia
  Interventions: Other: ePneumonia CDS
- Usual care: ED patients with pneumonia receiving usual care without electronic CDS

INTERVENTIONS:
Other: ePneumonia CDS — ePneumonia clinical decision support system for community-onset pneumonia
  Groups: ED Patients treated using ePneumonia CDS

SUMMARY:
The investigators plan to further develop a prototype, evidence-based, electronic clinical decision support system (CDSS) for pneumonia care (ePneumonia) with interoperability across Electronic Health Records in order to improve clinical outcomes and reduce healthcare resource utilization. The specific aims of this study are to evaluate the usability of ePneumonia adapted for Cerner and its impact on clinical, patient-centered and healthcare resource utilization outcomes in a stepped-wedge implementation study in 16 hospital emergency departments (EDs) across the Intermountain Healthcare integrated health system.

DETAILED DESCRIPTION:
Since the launch of a paper-based pneumonia care process model in 1994, decision support for pneumonia care has been under continuous development at Intermountain. Studies published in 2001 and 2006 demonstrated decreased mortality using paper-based methods. An electronic pneumonia Clinical Decision Support System was later developed in the original Intermountain computing environment and implemented in 4 regional emergency departments (ED) in 2011. This tool featured a novel mortality predictor and real-time synthesis of clinical data to guide diagnosis, risk stratification, admission triage and guideline-concordant treatment. An outcome study published in 2015 demonstrated reduction in mortality with tool use compared to usual care. Most recently, Intermountain researchers led by study co-Investigator, Dr. Brandon Webb, developed an innovative tool to predict risk of drug-resistant bacteria and demonstrated its potential to improve antibiotic use and outcomes.

The investigators have entered a robust phase of additional development and adaptation of ePneumonia into the Cerner Electronic Health Record (EHR) system. The objective of this study is to advance development of an evidence-based, electronic CDSS for pneumonia care with interoperability across EHRs in order to improve clinical outcomes and reduce healthcare resource utilization. The specific aim of this study is to evaluate the usability of ePneumonia and its associated impact on clinical, patient-centered and healthcare resource utilization outcomes in a stepped-wedge implementation study in 16 hospital EDs in the Intermountain Healthcare integrated health system.

* Hypothesis #1: Healthcare providers will affirm ePneumonia usability, lack of interference with clinical workflow and only minor unintended consequences of use.
* Hypothesis #2: In patients with community-onset pneumonia, ePneumonia use will improve clinical and patient-centered outcomes and decrease healthcare resource utilization.

One year of baseline clinical outcome data will be gathered for all 16 emergency departments. The first of 6 clusters of ED's will begin prospective data collection in January 2018, with the remaining coming on at 2 month intervals until ePneumonia has been deployed at all sites. An additional 1 year of data collection will be continued through 2019.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years who are identified by either (2a) ICD-10 codes for pneumonia; or acute respiratory failure or sepsis with secondary pneumonia codes or (2b) clinician completion of ePneumonia for Cerner.
* Intermountain Healthcare physicians working in the 16 ED's

Exclusion Criteria:

* Patients without radiographic confirmation of pneumonia
* subsequent episodes of pneumonia within the study period, so as not to over-represent patients with recurrent pneumonia caused by recurrent aspiration or structural lung disease, and
* immunosuppressed patients, such as those with AIDS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (1) All patients ≥ 18 years who are identified by either (2a) ICD-10 codes for pneumonia; or acute respiratory failure or sepsis with secondary pneumonia codes or (2b) clinician completion of ePneumonia for Cerner.
  Intermountain Healthcare physicians
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
30 day all-cause mortality | 30 days
  mortality within 30 days of initial ED visit

SECONDARY OUTCOMES:
Matching of patient disposition from the ED with ePneumonia recommendation | End of initial ED visit, <24 hours after ED arrival
  ePneumonia use will increase simple agreement between patient disposition from the ED with ePneumonia recommendation based on illness severity
Accuracy of Drug Resistance in Pneumonia (DRIP) score within the ePneumonia logic to predict Multi-Drug Resistant (MDR) pathogens | 30 days
  Sensitivity, specificity, positive and negative predictive values for DRIP score versus identified pathogens
Antibiotic utilization rates, in terms of appropriateness of spectrum | 30 days
  Antibiotic utilization rates, in terms of appropriateness of spectrum versus identified pneumonia pathogen
Rate of secondary hospital admission within 7 days for ED patients whose initial disposition was outpatient care | 7 days
  Rate of secondary hospital admission within 7 days for ED patients whose initial disposition was outpatient care
Direct costs | Duration of hospital stay, censored at 90 days
  ePneumonia use will produce lower direct costs (total and variable)
Length of stay | Duration of hospital stay, censored at 90 days
  ePneumonia use will shorten length of stay measured in hours
Healthcare providers will affirm ePneumonia usability, lack of interference with clinical workflow and only minor unintended consequences of use | 3 year study duration
  Qualitative outcome based on provider surveys

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Dean, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (17):
- United States (17):
  - Cassia Regional Hospital, Burley, Idaho
  - American Fork Hospital, American Fork, Utah
  - Cedar City Hospital, Cedar City, Utah
  - Delta Community Hospital, Delta, Utah
  - Fillmore Hospital, Fillmore, Utah
  - Heber Valley Hospital, Heber City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Sanpete Valley Hospital, Mount Pleasant, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Orem Community Hospital, Orem, Utah
  - Garfield Memorial Hospital, Panguitch, Utah
  - Park City Medical Center, Park City, Utah
  - Utah Valley Hospital, Provo, Utah
  - Sevier Valley Hospital, Richfield, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Bear River Hospital, Tremonton, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dean NC, Vines CG, Carr JR, Rubin JG, Webb BJ, Jacobs JR, Butler AM, Lee J, Jephson AR, Jenson N, Walker M, Brown SM, Irvin JA, Lungren MP, Allen TL. A Pragmatic, Stepped-Wedge, Cluster-controlled Clinical Trial of Real-Time Pneumonia Clinical Decision Support. Am J Respir Crit Care Med. 2022 Jun 1;205(11):1330-1336. doi: 10.1164/rccm.202109-2092OC. PMID 35258444